CLINICAL TRIAL: NCT05566964
Title: Descriptive Analysis of Real-world Data Collected with the ME&MGopen Mobile Application Developed for Myasthenia Gravis Patients
Brief Title: Descriptive Analysis of Real-world Data Collected with ME&MGopen
Status: Completed | Type: Observational
Sponsor: Ad scientiam (Other)
Responsible Party: Sponsor
Other Study IDs: ME&MGopen
Record Dates: First submitted 2022-09-07; First posted 2022-10-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ME&MGopen: Use of ME&MGopen mobile app, at home for 12 months
  Interventions: Device: ME&MGopen smartphone application

INTERVENTIONS:
Device: ME&MGopen smartphone application — Smartphone application includes digital tests and e-questionnaires

SUMMARY:
The ME&MGopen smartphone application is an investigational software for research purposes only, developed by Ad Scientiam. It features digital tests to assess the respiratory capacity ("My Breathing" Test), dysarthria ("My Voice" Test), ptosis ("My eyelids" test), as well as upper and lower limb muscle function ("My arms" Test and "My legs" Test). The mobile app also includes e-questionnaires related to activities of daily living, pain, insomnia, quality of life and depression. The objectives of the study are to collect data on patients' symptoms with the application in a real life setting, to assess adherence to the use of the tool, user experience and satisfaction with the application, and safety of use.

DETAILED DESCRIPTION:
The ME&MGopen smartphone application is an investigational software for research purposes only, developed by Ad Scientiam. It features digital tests to assess the respiratory capacity ("My Breathing" Test), dysarthria ("My Voice" Test), ptosis ("My eyelids" test), as well as upper and lower limb muscle function ("My arms" Test and "My legs" Test). The mobile app also includes e-questionnaires related to activities of daily living, pain, insomnia, quality of life and depression.

The objectives of the study are to collect data on patients' symptoms with the application in a real life setting, to assess adherence to the use of the tool, user experience and satisfaction with the application, and safety of use.

Analyses will also be performed to identify factors that may influence these parameters and provide levers for understanding and improvement. The existence of a possible learning effect on active testing will also be explored as a data point of interest.

The results will allow researchers to extend their knowledge of gMG from real-life data and of the use of digital tools in a gMG patient population

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 + years old
* Diagnosis of gMG with positive serologic test for anti-AChR autoantibody at screening
* Who has read the information sheet and signed the informed consent form
* Owns a personal smartphone which version is above 14 for IOS and 8 for Android included
* Able to use a smartphone
* Able to perform the ME&MG tests (based on investigator's judgment)
* Able to read language in which the mobile application is available (English, Spanish, German) and able to understand pictograms

Exclusion Criteria:

* Participating in another ME&MG trial
* Aged 17 years or younger
* A medical, psychological, or behavioral condition which interferes with compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living with generalized Myasthenia Gravis in the US and in Canada
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
To describe real-life upper limb weakness mesurements | Through study completion, an average of 12 months
  Time in seconds measured with the ME&MGopen smartphone application (holding the phone in one arm for as long as possible)
To describe real-life lower limb weakness measurements | Through study completion, an average of 12 months
  Number of sit-to-stand actions measured with the ME&MGopen smartphone application (1 minute sit-to-stand test)
To describe real-life ptosis measurements | Through study completion, an average of 12 months
  Margin-Reflex Distance 1 (MRD1) measured with the ME&MGopen smartphone application
To describe real-life dysarthria measurements | Through study completion, an average of 12 months
  Time in seconds measured with the ME&MGopen smartphone application
To describe real-life respiratory capacity measurements | Through study completion, an average of 12 months
  Time in seconds measured with the ME&MGopen smartphone application : saying "aaaaahhh" for as long as possible
To describe activities of daily living | Through study completion, an average of 12 months
  Myasthenia Gravis Activities of Daily Living scores (0-24) higher score meaning a worse outcome
To describe depression symptoms | Through study completion, an average of 12 months
  Patient Health Questionnaire-8 (0-12) higher score meaning a worse outcome
To describe pain symptoms | Through study completion, an average of 12 months
  Pain Likert scale scores(0-10) higher score meaning a worse outcome
To describe insomnia symptoms | Through study completion, an average of 12 months
  Insomnia Severity Index scores (0-28) higher score meaning a worse outcome, 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
To describe quality of life related to MG | Through study completion, an average of 12 months
  Myasthenia Gravis Quality of Life 15-item Scale revised scores (0-30) higher score meaning a worse outcome
To describe quality of life | Through study completion, an average of 12 months
  36-Item Short Form Survey version 1 (0-100) higher score meaning a better outcome

SECONDARY OUTCOMES:
To evaluate the reliability of the digital tests performed at home in real-life | Baseline, month 1, month 2, month 3, Month 4, month 5, month 6, month 7, month 8, month 9, month 10, month 11, month 12
  The intraclass correlation coefficient mean k raters (ICCk; k=month) will be used to assess the monthly reliability at home of digital tests from the beginning to the end of participation :
  At-home MET At-home MBT At-home MVT At-home MAT At-home MLT
To assess adherence to the mobile application | through study completion, 30 months
  Descriptive analysis of the mobile application's adherence data (number of completed questionnaires, carried tests, number of sessions performed etc.)
To assess the satisfaction and user experience with the smartphone application | through study completion, 30 months
  Descriptive analysis (counts/percentages) of the answers to the user experience and satisfaction questionnaires related to the use of the ME&MGopen smartphone application
To assess user behavior | through study completion, 30 months
  Description of user behavior (counts/percentages)
To assess safety of use of the smartphone application | through study completion, 30 months
  Descriptive analysis of adverse events (AEs) related and unrelated to the use of the application. Adverse event data will be reported in a table and expressed as number and percentage, differentiating mild, moderate and severe AEs.
To evaluate the effect of different frequencies of assessments of the digitals tests on the onset of learning effect | through study completion, 30 months
  p-value
To analyze correlations between digital tests, e-questionnaires, socio demographic data, treatments | through study completion, 30 months
  Matrix correlation to estimate Pearson's correlation coefficient for each pair of relevant variables.
To evaluate the ability of the Health Belief Model to predict user behavior towards the smartphone application | through study completion, 30 months
  coefficient of correlation between dimensions of the Health Belief Model and device use
To identify if socio-demographic data, treatment status, severity, satisfaction and user experience could influence the results to the digital tests and questionnaires | through study completion, 30 months
  p-value from multiple regression
To identify if socio-demographic data, treatment status, severity, satisfaction and user experience could influence the reliability of the digital tests | through study completion, 30 months
  p-value from multiple regression
To identify if depression , activities of daily living and satisfaction could influence the adherence to the smartphone application | through study completion, 30 months
  p-value from multiple regression
To identify if socio-demographic data or treatment status could influence satisfaction with the smartphone application | through study completion, 30 months
  p-value from multiple regression
To explore the existing association between the ME&MG tests scores obtained at home and the results labeled by a trained evaluator | through study completion, 30 months
  coefficient of correlation

CONTACTS AND LOCATIONS:
Locations (3):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States
- University Health Network, Toronto, Ontario, Canada
- Lindus Health, London, Greater london, United Kingdom

IPD SHARING:
Plan to Share IPD: No